CLINICAL TRIAL: NCT03154125
Title: A Study to Evaluate the Effectiveness, Pharmacokinetics, Safety, and Acceptability of Sayana® Press When Injected Every Four Months
Brief Title: Sayana® Press Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 926400
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Results first posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Contraception
MeSH Terms: interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Intervention Model Description: All participants will receive the same study drug, Sayana® Press. However, women will be randomized to receive their injections in the abdomen, back of the upper arm, or upper thigh to control for potential confounding when assessing relationships between SC injection site, efficacy, and PK. One cohort of N=630 women will be randomized 1:1 to receive their injections in the abdomen or thigh, and a separate PK cohort of N=120 women agreeing to MPA testing will be randomized 1:1:1 to receive their injections in the abdomen, upper thigh, or back of the upper arm. Randomization will be stratified by cohort and site using appropriate randomly permuted block sizes.
Who Masked: Outcomes Assessor
Masking Description: Neither participants nor site staff will be blinded to SC injection sites. However, laboratory staff analyzing serum MPA specimens and staff at FHI 360 responsible for adjudicating pregnancy outcomes and coding adverse events will be blinded to individual participant injection site assignments for the duration of each participant's follow up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Abdomen (Experimental): Sayana® Press (MPA injectable suspension, 104 mg/0.65 mL, pre-filled in the UnijectTM delivery injection system) injected subcutaneously every 4 months (17-18 weeks) for 3 treatment cycles (12 months).
  Interventions: Drug: Sayana® Press
- Upper thigh (Experimental): Sayana® Press (MPA injectable suspension, 104 mg/0.65 mL, pre-filled in the UnijectTM delivery injection system) injected subcutaneously every 4 months (17-18 weeks) for 3 treatment cycles (12 months).
  Interventions: Drug: Sayana® Press
- Back of the upper arm (Experimental): Sayana® Press (MPA injectable suspension, 104 mg/0.65 mL, pre-filled in the UnijectTM delivery injection system) injected subcutaneously every 4 months (17-18 weeks) for 3 treatment cycles (12 months).
  Interventions: Drug: Sayana® Press

INTERVENTIONS:
Drug: Sayana® Press — The active ingredient in Sayana® Press is Medroxyprogesterone acetate (MPA). Sayana® Press (MPA injectable suspension, 104 mg/0.65 mL, pre-filled in the UnijectTM delivery injection system) for subcutaneous injection.
  Other Names: medroxyprogesterone acetate (MPA) injectable suspension

SUMMARY:
This is a randomized clinical trial designed to evaluate the effectiveness, safety and acceptability of Sayana® Press when injected every 4 months (17-18 weeks) for 3 treatment cycles (12 months) of use.

DETAILED DESCRIPTION:
This is a randomized, partially-blinded, multi-center, parallel-group study to evaluate the effectiveness, PK, safety, and acceptability of Sayana® Press when injected every 4 months (17-18 weeks) rather than the currently prescribed 3-month (12-14 weeks) regimen.

A total of 750 healthy, sexually active women aged 18 to 35 years with regular menstrual cycles and no DMPA use in the previous 12 months will be enrolled and followed for pregnancy. Among all enrolled, 710 will be randomized to receive injections in the abdomen or upper thigh in accordance with the PATH Sayana® injection instructions, which are consistent with prescribing information, for the primary effectiveness analysis. An additional 40 women will be randomized to receive injections subcutaneously in the back of the upper arm to assess whether differences in PK may exist which could impact the grace period for reinjections for that injection site.

A single MPA serum sample will be collected from all participants at baseline. All participants will receive re-injections at month 4 and month 8, and complete their scheduled follow-up at month 12. There will be a plus 7-day grace period for re-injections, but women who are up to 28 days late may continue treatment if they have a negative urine pregnancy test. Urine pregnancy testing will be performed at month 4, at study exit and at any other time during the study if clinically indicated. Participants will be evaluated for injection site reactions and asked to provide information on adverse events, prohibited concomitant medication and other contraceptive use, vaginal bleeding, and method acceptability at all regular follow-up visits (i.e., not including the PK visits at Months 2 and 3). Serious adverse events and adverse events leading to product withdrawal, will be recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* not pregnant and no desire to become pregnant in the next 18 months
* regular menstrual cycles (25 to 35 days in length when not using hormonal contraception, pregnant, or lactating)
* at risk of pregnancy (no diagnosis of infertility, no history of tubal ligation or hysterectomy, and an average of 1 or more unprotected acts of vaginal intercourse per month)
* in good general health as determined by a medical history
* 18 to 35 years of age, inclusive
* willing to provide informed consent, follow all study requirements, and rely on Sayana® Press injected every 4 months as the only means of contraception for 12 months
* has only one sexual partner and expects to have that same sexual partner for the next 12 months

Exclusion Criteria:

* has a primary partner who has received a vasectomy or is otherwise sterile
* medical contraindications to depot medroxyprogesterone acetate (DMPA) per World Health Organization medical eligibility criteria for contraceptive use
* known HIV-infection (for her or her partner)
* diagnosis or treatment for a sexually transmitted infection in the past month (for her or a partner), excluding recurrent herpes or condyloma
* received an injection of a progestin-only containing contraceptive (DMPA or norethisterone enanthate) in the past 12 months
* received an injection of a combined injectable contraceptive in the past 6 months
* known or suspected allergic reaction to DMPA
* used a levonorgestrel-releasing intrauterine system, NuvaRing, contraceptive patch, oral contraceptives or a contraceptive implant in the 7 days prior to enrollment (PK cohort only)
* previous (within 1 month prior to enrollment), current or planned (in the next 12 months) use of an investigational drug, prohibited drug per protocol or other drug which in the opinion of the site investigator could complicate study findings
* has been pregnant in the past month
* is lactating
* plans to move to another location in the next 12 months
* has a social or medical condition which in the opinion of the site investigator would make study participation unsafe, or interfere with adherence to protocol requirements.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 750 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vera Halpern, MD, Study Director — FHI 360
Locations (3):
- Universidade Estadual de Campinas (UNICAMP), Campinas, Brazil
- Instituto Chileno De Medicina Reproductiva (ICMER), Santiago, Chile
- Asociación Dominicana Pro Bienestar de la Familia, Inc. (PROFAMILIA), Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: Yes
Study sites will collect baseline and longitudinal data among 750 women in Brazil, Chile and the Dominican Republic relevant to the protocol objectives including demographics; sexual, reproductive and medical history; acceptability; serious adverse events; concomitant medication use and laboratory data (including serum blood medroxyprogesterone acetate concentrations in a subset of women).
  • FHI 360 will submit the study dataset using the platform-independent and non-proprietary comma separated values (also known as [CSV]) format. The study dataset will be posted to a third-party data repository, then the link will be submitted to USAID's Data Development Library within 30 calendar days after the dataset is first used to produce an Intellectual Work.
  A code book defining all variables, a data dictionary describing the relationships among the files within the dataset, and a document describing the methodology used to collect the data will be shared with the study dataset.
Time Frame: Within 30 calendar days after the dataset is first used to produce an Intellectual Work

REFERENCES:
- [Derived] Burke HM, Packer C, Fuchs R, Brache V, Bahamondes L, Salinas A, Veiga N, Miller A, Deese J. Acceptability of the contraceptive Sayana(R) Press when injected every four months: Results from a twelve-month trial in Brazil, Chile and the Dominican Republic. Contraception. 2022 Sep;113:95-100. doi: 10.1016/j.contraception.2022.04.007. Epub 2022 Apr 26. PMID 35483431
- [Derived] Deese J, Brache V, Bahamondes L, Salinas A, Jorge A, Veiga N Jr, Fuchs R, Miller A, Taylor D, Halpern V, Dorflinger L. Contraceptive effectiveness, pharmacokinetics, and safety of Sayana(R) Press when injected every four months: a multicenter phase 3 trial. EClinicalMedicine. 2022 Jan 29;44:101273. doi: 10.1016/j.eclinm.2022.101273. eCollection 2022 Feb. PMID 35128365

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 836 Screened, 86 Not Enrolled - Medically Ineligible: 26, Declined to Enroll: 24, Ineligible due to Sexual Behavior or Recent Contraceptive Use: 19, Unable to Comply with Study Req.:15, Investigator Discretion: 2
Period: Overall Study
Arm/Group | Abdomen | Upper Thigh | Back of the Upper Arm
Started | 355 | 355 | 40
Randomized to PK Cohort | 40 | 40 | 40
PK Population | 35 | 33 | 32
Excluded From PK Population | 5 | 7 | 8
Completed | 279 | 278 | 32
Not Completed | 76 | 77 | 8
Not completed — Lost to Follow-up | 11 | 11 | 0
Not completed — Withdrawal by Subject | 49 | 55 | 8
Not completed — Physician Decision | 13 | 6 | 0
Not completed — Protocol Violation | 3 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abdomen | Upper Thigh | Back of the Upper Arm | Total
Number analyzed (Participants) | 355 | 355 | 40 | 750
Age, Customized [Count of Participants; unit: Participants]
  participants18-29 years | 266 | 273 | 31 | 570
  participants 30-40 years | 89 | 82 | 9 | 180
Sex/Gender, Customized [Number; unit: participants]
  Female | 355 | 355 | 40 | 750
Race/Ethnicity, Customized [Number; unit: participants]
  White | 104 | 104 | 20 | 228
  Black | 28 | 29 | 1 | 58
  Bi-/Multi-racial | 223 | 222 | 19 | 464
Education [Count of Participants; unit: Participants]
  Participants ≤9 years | 94 | 91 | 7 | 192
  Participants >9 years | 261 | 264 | 33 | 558
Average times have vaginal sex per month with male partner [Mean (Standard Deviation); unit: Events per month] | 12.1 (7.27) | 11.9 (8.09) | 10.2 (6.23) | 11.9 (7.62)
Weight [Mean (Standard Deviation); unit: kg] | 72.7 (18.72) | 71.1 (16.89) | 72.1 (15.21) | 71.9 (17.70)
Height [Mean (Standard Deviation); unit: cm] | 160.7 (5.98) | 160.5 (6.70) | 160.6 (6.38) | 160.6 (6.34)

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Pregnancy
Description: Pregnancy is defined as having a positive urine pregnancy test. Positive urine tests will be confirmed by ultrasound and/or serum hCG testing whenever possible. The primary efficacy analysis will be based on the pregnancy Pearl Index, computed as the number of pregnancies that occur during the treatment period multiplied by 100 and divided by the number of WY of treatment contributed to the Treated Analysis Set among women receiving injections in the abdomen or thigh.
Time Frame: 12 months after treatment initiation
Population: The primary study objective is to evaluate the effectiveness of Sayana® Press when injected subcutaneously every 4 months among women in the Treated Analysis set who received injections in the abdomen or upper thigh. This outcome measure was pre-specified to only assess participants who were injected in the abdomen and upper thigh.
Measure: Number (95% Confidence Interval); unit: Pregnancies per 100 women years
Arm/Group | Abdomen | Upper Thigh
Number analyzed (Participants) | 355 | 355
Pregnancies per 100 women years | 0 [0 to 1.18] | 0 [0 to 1.17]

2. Secondary Outcome: Serum MPA Concentrations in a Subset of 120 Participants
Description: Pharmacokinetic endpoints include serum MPA concentrations at month 2, 3, 4, 8, and 12.
Time Frame: 2, 3, 4, 8, and 12 months after treatment initiation
Population: Subset of study participants consenting to MPA concentration analysis. Excluding participants who did not contribute blood specimens, who had baseline MPA >0.05 ng/mL, or who required the use of more than 1 Sayana Press unit or their baseline injection. Also, the analysis set excludes any MPA specimens collected during a time when a participant reports using a concomitant medication that may impact the PK of MPA. The analysis set excludes any MPA results after an injection with more than 1 unit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Abdomen | Upper Thigh | Back of the Upper Arm
Number analyzed (Participants) | 35 | 33 | 32
ng/mL
  Trough concentration at Month 2: number analyzed (Participants) | 34 | 32 | 31
  Trough concentration at Month 2 | 0.503 (0.263) | 0.355 (0.155) | 0.490 (0.264)
  Trough concentration at Month 3: number analyzed (Participants) | 34 | 31 | 31
  Trough concentration at Month 3 | 0.367 (0.145) | 0.328 (0.160) | 0.337 (0.180)
  Trough concentration at Month 4: number analyzed (Participants) | 33 | 31 | 31
  Trough concentration at Month 4 | 0.299 (0.131) | 0.267 (0.133) | 0.248 (0.105)
  Trough concentration at Month 8: number analyzed (Participants) | 30 | 27 | 25
  Trough concentration at Month 8 | 0.455 (0.159) | 0.404 (0.145) | 0.305 (0.125)
  Trough concentration at Month 12: number analyzed (Participants) | 29 | 22 | 22
  Trough concentration at Month 12 | 0.502 (0.148) | 0.431 (0.127) | 0.362 (0.155)

3. Secondary Outcome: Occurrence of Serious Adverse Events (SAEs) and Adverse Events (AEs) Leading to Product Withdrawal
Description: The overall safety of study drug will be assessed throughout the study by evaluating the occurrence of SAEs and AEs leading to product discontinuation, blood pressure and weight at regularly scheduled visits, and changes in bleeding pattern.
Time Frame: 12 months after treatment initiation
Population: Whole study population
Measure: Number; unit: Events
Units Other Than Participants: Events
Groups:
- Abdomen; Upper Thigh; Back of Upper Arm: Total count of SAEs and AEs, AEs leading to withdrawal, and AEs which are grade 1 or higher
Arm/Group | Abdomen | Upper Thigh | Back of Upper Arm
Number analyzed (Participants) | 355 | 355 | 40
Number analyzed (Events) | 34 | 38 | 5
Events
  Abdominal pain lower | 0 | 2 | 0
  Injection site discolouration | 1 | 0 | 0
  Injection site oedema | 0 | 1 | 0
  Injection site reaction | 9 | 6 | 0
  Lower limb fracture | 1 | 0 | 0
  Weight decreased | 1 | 3 | 0
  Weight increased | 2 | 0 | 1
  Pain in extremity | 0 | 1 | 0
  Cerebrovascular accident | 1 | 0 | 0
  Headache | 1 | 1 | 0
  Libido decreased | 2 | 0 | 0
  Mood altered | 1 | 0 | 0
  Amenorrhoea | 2 | 5 | 0
  Menometrorrhagia | 0 | 1 | 0
  Menstruation irregular | 9 | 14 | 4
  Metrorrhagia | 0 | 2 | 0
  Oligomenorrhoea | 1 | 1 | 0
  Pelvic pain | 1 | 0 | 0
  Vulvovaginal dryness | 0 | 1 | 0
  Acne | 2 | 0 | 0

4. Secondary Outcome: Acceptability of Sayana® Press
Description: Perception of bleeding patterns and other responses to acceptability questions will be summarized using descriptive statistics based on routine questions asked at regularly scheduled visits (enrollment, months 4 and 8, and final). Acceptability data collected during unscheduled visits are not included in this table.
Time Frame: 12 months after treatment initiation
Population: Treated Population: Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- Abdomen: Study Participants Receiving Injections in Abdomen and Completing Final Visit. Participants Not Included: 11 LTF, 16 Early Discontinuation
- Upper Thigh: Study Participants Receiving Injections in Upper Thigh and Completing Final Visit. Participants Not Included: 11 LTF, 8 Early Discontinuation
- Back of Upper Arm: Study Participants Receiving Injections in Back of Upper Arm and Completing Final Visit. Participants Not Included: 2 Early Discontinuation
Arm/Group | Abdomen | Upper Thigh | Back of Upper Arm
Number analyzed (Participants) | 328 | 336 | 38
Participants
  Would you like to use Sayana Press as a 4-month method in the future if proven effective? : Yes | 306 | 313 | 34
  Would you like to use Sayana Press as a 4-month method in the future if proven effective? : No | 22 | 23 | 4

5. Other Pre Specified Outcome: Return to Ovulation After 12 Months of Use of Sayana Press When Injected Every Four Months.
Description: Return to ovulation among a subset of study participants who received month 4 and month 8 injections and plan to use non-hormonal methods of contraception, or no contraception for up to a maximum of 12 months from the last study injection. Ovulation is defined as a single elevated serum progesterone (P ≥4.7 ng/mL) or a confirmed pregnancy test.
Time Frame: A maximum of 12 months from the last study injection.
Population: A subset of ~20 participants at study sites in Brazil and Dominican Republic who received month 4 and month 8 injections and planned to use a non-hormonal contraceptive method, or no contraception, after study discontinuation. One participant who received an injection in the abdomen discontinued early and was censored from analysis at 41 weeks past final injection. The subset was restricted to participants included in the primary analysis, those injected in the abdomen or thigh.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abdomen | Upper Thigh
Number analyzed (Participants) | 8 | 11
Percentage of participants
  Women who ovulated or became pregnant by 42 weeks after final injection | 25 [3.2 to 65.1] | 18.2 [2.3 to 51.8]
  Women who ovulated or became pregnant by 50 weeks after final injection | 50 [15.7 to 84.3] | 54.5 [23.4 to 83.3]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Abdomen | Upper Thigh | Back of the Upper Arm
All-Cause Mortality (participants affected / at risk) | 0/355 | 0/355 | 0/40
Serious Adverse Events (participants affected / at risk) | 2/355 | 0/355 | 0/40
Other Adverse Events (participants affected / at risk) | 32/355 | 38/355 | 5/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abdomen (N=355) | Upper Thigh (N=355) | Back of the Upper Arm (N=40)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abdomen (N=355) | Upper Thigh (N=355) | Back of the Upper Arm (N=40)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 2 | 0
Injection Site Discolouration (General disorders) | 1 | 0 | 0
Injection Site Oedema (General disorders) | 0 | 1 | 0
Injection Site Reaction (General disorders) | 9 | 6 | 0
Weight Decreased (Investigations) | 1 | 3 | 0
Weight Increased (Investigations) | 2 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 0
Libido Decreased (Psychiatric disorders) | 2 | 0 | 0
Mood Altered (Psychiatric disorders) | 1 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 2 | 5 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Menstruation Irregular (Reproductive system and breast disorders) | 9 | 14 | 4
Metrorrhagia (Reproductive system and breast disorders) | 0 | 2 | 0
Oligomenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal Dryness (Reproductive system and breast disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT03154125/Prot_001.pdf
  • Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/25/NCT03154125/SAP_002.pdf
  • Informed Consent Form (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT03154125/ICF_000.pdf